CLINICAL TRIAL: NCT06982144
Title: AI-based Prediction Model of Difficult Tracheal Intubation Using Medical Image Parameters
Status: Not yet recruiting | Type: Observational
Sponsor: Mu Dong Liang (Other)
Responsible Party: Sponsor-Investigator, Mu Dong Liang, Professor, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: 2025R-0037
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Difficult Airway
Keywords: difficult airway; AI-based method; medical imaging; prediction model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients scheduled for selective surgery

SUMMARY:
Difficult airway is a life-threatening event during anesthesia. Prediction model is helpful to detect high-risk patients and decrease the risk of un-anticipated difficult airway. Present models are usually based on Mallampati grade and the width of mouth open. However, the prediction accuracy is only about 0.7-0.8 in different populations. Present study is designed to investigate if AI-based prediction model using medical imaging parameters (such as CT and MRI) can increase the accuracy of prediction model.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years old;
2. surgical patients undergoing general anesthesia with endotracheal intubation;
3. with head and neck CT examination results
4. Consent to participate in the study.

Exclusion Criteria:

1. The presence of laryngeal edema;
2. The presence of airway stenosis, including internal airway stenosis (such as foreign body or tumor) or stenosis caused by external tracheal mass compression;
3. tracheo-esophageal fistula;
4. severe gastroesophageal reflux;
5. previous upper airway surgery, such as laryngeal cancer radical surgery, snoring surgery, etc.

6）participating in other research projects

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck CT data undergoing surgery under general anesthesia with endotracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 228 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
The accuracy of prediction model based on AI analysis of medical imaging parameters | day 1 (From enrollment to the end of anesthesia induction)
  To establish a prediction model for difficult tracheal intubation based on medical imaging parameters (such as CT and MRI) using AI algorithms and verify its predictive accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No